CLINICAL TRIAL: NCT05886608
Title: Evaluation of the Effect of the AI500™ SINGLE-DOSE GEL Medical Device in Patients With Reduced Knee Function: a Post-market Confirmatory Interventional, Single Arm Clinical Investigation
Brief Title: Evaluation of the Effect of the AI500™ SINGLE-DOSE GEL Medical Device in Patients With Reduced Knee Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Contrad Swiss SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTD-SW AI500 2021
Record Dates: First submitted 2023-05-12; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Pain, Acute; Pain, Chronic; Knee Injuries; Knee Osteoarthritis; Knee Arthritis; Knee Pain Swelling
Keywords: Knee; Pain; Hyaluronic Acid; Peptides; Non-invasive
MeSH Terms: conditions — Acute Pain; Chronic Pain; Knee Injuries; Osteoarthritis, Knee; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AI500 single-dose gel (Other): Interventional study on AI500 1.5 mL will be topically administered twice: the first at T0 and the second 24h from T0
  Interventions: Device: AI 500™ SINGLE-DOSE GEL

INTERVENTIONS:
Device: AI 500™ SINGLE-DOSE GEL — AI500™ SINGLE-DOSE GEL is a hydrogel to be applied to intact skin, intended to provide relief in cases of pain due to tension in muscles and adjacent tissues, to improve movement and function.

SUMMARY:
Evaluation of the effect of the AI500™ SINGLE-DOSE GEL medical device in patients with reduced knee function

DETAILED DESCRIPTION:
The aim of this post-market confirmatory interventional clinical investigation is to evaluate the performance and safety of AI500™ SINGLE-DOSE GEL in patients with reduced knee function.

ELIGIBILITY:
Inclusion Criteria:

1. Signed patient informed consent form (ICF).
2. Male or Female aged ≥ 18 years at the time of the signature of ICF.
3. Presenting with reduced knee function caused by osteoarthritis flare-ups, meniscal injuries, ligament injuries, inflammation of soft tissues, assessed as 20-45 rating according to the WOMAC function scale.
4. Willingness to follow all study procedures, including attending all site visits, tests, and examinations.
5. Willingness to follow indications.

Exclusion Criteria:

1. Use of analgesics within the 24 hours prior to V0.
2. Damaged, infected, or ulcerated skin in the area of treatment.
3. Ongoing cutaneous allergies.
4. Serious and chronic pathological skin conditions (i.e., rosacea, psoriasis, vitiligo) or lesions including cancer with/without ongoing antitumor therapy.
5. Patients suffering from muscular dystrophy.
6. Patients presenting with bone fractures or severe injuries (including locked knee).
7. Severely disabled arthritic patients using a wheelchair.
8. Allergy to device components (Sodium hyaluronate; SHPolypeptide- 6; Glycerin; Propylene glycol; Ethylhexylglycerin; Panthenol; PEG-40 hydrogenated castor oil; Sodium hydroxide; Xanthan gum; Phenoxyethanol; Benzoic Acid; Carbomer; Dehydroacetic Acid; Disodium EDTA).
9. Immune system illnesses.
10. Uncontrolled systemic diseases.
11. Known drug and/or alcohol abuse.
12. Mental incapacity that precludes adequate understanding or cooperation.
13. Participation in another investigational study.
14. Pregnancy or breastfeeding.
15. Patients with both knees affected/damaged.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-03-16 (Actual)

PRIMARY OUTCOMES:
Clinical performance of AI500™ SINGLE DOSE GEL in improving knee function after 1 week | 1 Week
  To evaluate the clinical performance of AI500™ SINGLE DOSE GEL in improving knee function after 1 week of treatment, change from baseline (V0) to week 1 (V3) in Western Ontario and McMasters Universities Osteoarthritis Index (WOMAC) Physical Function score will be evaluated.
  The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function.

SECONDARY OUTCOMES:
Clinical performance of AI500™ SINGLE DOSE GEL in improving knee function after 48 hours | 2 days
  To evaluate the clinical performance of AI500™ SINGLE DOSE GEL in improving knee function after 48 hours of treatment, change from baseline to 48 hours (V2) in WOMAC Physical Function score will be evaluated.
  The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function.
Clinical performance of AI500™ SINGLE DOSE GEL in alleviating pain after 24h and 48h of treatment. | 2 days
  To evaluate the clinical performance of AI500™ SINGLE DOSE GEL in alleviating pain after 24h and 48h of treatment, change in NRS between V0 and V1, and between V0 and V2 will be analysed.
  NRS Score has a range of 0-10 for pain; 0=no pain; 10=max pain.
Safety and Tolerability of AI500™ SINGLE DOSE GEL | 1 week
  To evaluate the safety and tolerability of AI500™ SINGLE DOSE GEL, physical examination and adverse events (AEs), including of the relationship of the AE to the IP (e.g., local allergic reaction), will be assessed through the study.
  Safety and tolerability of the AI500™ will be evaluated through a the completion of a specific questionnaire by the patient, the five-points Likert scale in which 1 means Strongly disagree with the assertion and 5 means Strongly agree

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas Research Hospital, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: Undecided